CLINICAL TRIAL: NCT04823273
Title: Blood Transfusion Reduction Quality Improvement Project
Brief Title: Blood Transfusion Reduction - QI Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 19-0918
Record Dates: First submitted 2021-03-23; First posted 2021-03-30 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Blood Transfusion
Keywords: blood transfusion; EHR interventions; user-centered design; high-value care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- General improvement (Experimental): Using the expertise of the study personnel, electronic-health record system architects working for UCHealth, and incorporating feedback from the users who participated in the user-centered design sessions we made changes to the blood transfusion order-set as well as the "prepare" and "transfuse" orders. The intention of the changes to the interface are to be more intuitive for ordering clinicians.
  Interventions: Behavioral: General improvement
- In-line help text (Experimental): In addition to general improvement changes, subjects exposed to the in-line help text arm receive text detailing evidence-based transfusion recommendations that appear if the most recent hemoglobin level is above 7.0 g/dL. This text appears within the transfusion order but is non-interruptive as it does not require users to acknowledge the text nor does is require any additional keystrokes or clicks.
  Interventions: Behavioral: In-line help text
- Interruptive alert (Experimental): In addition to general improvement changes, subjects exposed to the interruptive alert arm receive text detailing evidence-based transfusion recommendations that appear if the most recent hemoglobin level is above 7.0 g/dL. In contrast to the in-line help text arm, this arm includes an interruptive alert that appears when the user selects the transfusion order. This alert offers users the option to remove the order which results in no-blood product ordered. Alternatively, users may continue to order blood and are asked to select the reason for proceeding with the intended order.
  Interventions: Behavioral: Interruptive alert

INTERVENTIONS:
Behavioral: General improvement — Changes to interface to be more intuitive.
  Arms: General improvement
Behavioral: In-line help text — General improvement + in-line help text
  Arms: In-line help text
Behavioral: Interruptive alert — General improvement + interruptive alert
  Arms: Interruptive alert

SUMMARY:
Blood Banks of large medical centers have large annual budgets, typically millions of dollars. Blood product wastage results in not only in a loss of the product's cost, but also of the fees involved in transporting, handling, and administering these products. Optimal utilization of blood products requires a balance between maximizing patient clinical outcomes while avoiding unnecessary costs and risks associated with transfusions. This project will specifically focus on packed red blood cell transfusions (pRBCs). There are clear guidelines for transfusing pRBCs however these guidelines are not always followed. pRBC transfusions outside of recommended guidelines is associated with increased risk of harm to patients.

Our aim is to improve adherence to guideline indicated pRBC transfusions for patient in the UCHealth system thereby decreasing inappropriate (non-guideline indicated) pRBC transfusions. We will conduct a QI project seeking to improve pRBC transfusion guideline adherence. This project will involve data review to establish baseline rates, multimodal interventions to improve adherence to pRBC transfusion guidelines including provider education, modifications to the electronic ordering interface, and changing blood back policies at participating institutions.

ELIGIBILITY:
Inclusion Criteria:

* All physicians and nurses with access to order inpatient blood transfusions through a hospital-based EMR.
* All physicians and nurses ordering blood for individuals over the age of 18.

Exclusion Criteria:

* All physicians and nurses ordering blood transfusion ordering blood in the OR
* Blood ordered through massive transfusion protocol

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1640 (Actual)
Dates: Start 2021-04-06 (Actual); Primary Completion 2022-04-05 (Actual); Study Completion 2022-10-15 (Actual)

PRIMARY OUTCOMES:
Blood Transfusion Orders | 78 weeks
  Number of patients who received blood transfusions during the study by arm.
Guideline Concordance Measured by Pre-Transfusion Hemoglobin Values Per Transfusion | 78 weeks
  The American Association of Blood Banks recommends a restrictive threshold of a pre-transfusion hemoglobin level of less than 7.0g/dL for the vast majority of inpatients. Transfusions with Hemoglobin levels above 7 will be compared in arm 1 vs 2 +3 combined; arm 2 vs arm 3.
Guideline Concordance Measured by Number of Units Ordered Per Transfusion | 78 weeks
  The American Association of Blood Banks recommends a restrictive threshold of a single unit pRBC transfusion for the vast majority of inpatients. This outcome will compare hemoglobin levels, units transfused in arm 1 verses arms 2 and 3 combined and arm 2 verses arm 3.

OTHER OUTCOMES:
Historical Blood Transfusion Orders | Baseline
  Number of patients who received blood transfusions during the 18 months prior to study start in the EHR at the same hospital.
Historical Guideline Concordance Measured by Pre-Transfusion Hemoglobin Values Per Transfusion | Baseline
  The American Association of Blood Banks recommends a restrictive threshold of a pre-transfusion hemoglobin level of less than 7.0g/dL for the vast majority of inpatients. Historical data for 18 months prior to study start will be collected from EHR records for transfusions orders placed for patients with Hemoglobin levels above 7.
Guideline Concordance Measured by Number of Units Ordered Per Transfusion | Baseline
  The American Association of Blood Banks recommends a restrictive threshold of a single unit pRBC transfusion for the vast majority of inpatients. Historical data for 18 months prior to study start will be collected from EHR records for the number of units transfused per blood transfusion order.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Ho, MD, PhD, Study Director — University of Colorado Denver Anschutz Medical Campus; Tyler Anstett, DO, Principal Investigator — University of Colorado Denver Anschutz Medical Campus
Locations (1):
- UCHealth University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mistry N, Richardson V, Carey E, Porter S, Pincus S, Novins-Montague S, Elmer M, Lin CT, Ho PM, Anstett T. General improvements versus interruptive or non-interruptive alerts in the blood order set: study protocol for a randomized control trial to improve packed red blood cell utilization. Trials. 2023 May 8;24(1):314. doi: 10.1186/s13063-023-07319-8. PMID 37158929